CLINICAL TRIAL: NCT03271411
Title: Extension of EMDR vs. PC For Motor Vehicle Accident Trauma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Trauma Institute & Child Trauma Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017-1002
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Trauma, Psychological; Motor Vehicle Accident
MeSH Terms: conditions — Psychological Trauma

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eye movement desensitization and reprocessing (EMDR) arm (Experimental)
  Interventions: Behavioral: EMDR-based Flash technique
- Progressive counting (PC) arm (Experimental)
  Interventions: Behavioral: PC-based Flash technique

INTERVENTIONS:
Behavioral: EMDR-based Flash technique — Initial EMDR session (with Flash technique) of up to three hours; about one week later, follow-up session of up to one hour
  Arms: Eye movement desensitization and reprocessing (EMDR) arm
Behavioral: PC-based Flash technique — Initial PC session (with Flash technique) of up to three hours; about one week later, follow-up session of up to one hour
  Arms: Progressive counting (PC) arm

SUMMARY:
This is an extension of a randomized clinical trial comparing eye movement desensitization and reprocessing (EMDR) to progressive counting (PC) for volunteers from the community who are distressed by the memory of a motor vehicle accident. The purpose of this extension is to add Phil Manfield's recently developed Flash technique as a precursor to both EMDR and PC, to see a) if that has any impact on participant retention, treatment effectiveness, or treatment efficiency; and b) if such impact is equivalent with EMDR and PC.

ELIGIBILITY:
Inclusion Criteria:

* adult reporting distress related to motor vehicle accident-related trauma
* English-speaking

Exclusion Criteria:

* already in therapy in which the memory of interest is being actively addressed with a structured/focused trauma resolution method
* any obvious/urgent need for more comprehensive psychotherapy (based on initial screening interview)
* any indication of instability during interactions prior to the therapy session
* an average score on the Dissociative Experiences Scale of 30 or greater, if (as per follow-up questions) indicating a likely dissociative disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2017-08-30 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in SUDS following treatment | Administered pre-treatment, two weeks post-treatment, and 12 weeks post-treatment
  Subjective Units of Distress Scale
Change in PRS following treatment | Administered pre-treatment, two weeks post-treatment, and 12 weeks post-treatment
  Problem Rating Scale
Change in PDS following treatment | Administered pre-treatment, two weeks post-treatment, and 12 weeks post-treatment
  PTSD Diagnostic Scale

CONTACTS AND LOCATIONS:
Overall Officials: Ricky Greenwald, PsyD, Principal Investigator — Trauma Institute & Child Trauma Institute
Locations (1):
- Trauma Institute & Child Trauma Institute, Northampton, Massachusetts, United States